CLINICAL TRIAL: NCT02341989
Title: A Randomized Phase III Study Comparing One Course of Adjuvant Bleomycin, Etoposide and Cisplatin (BEP) and One Course of Carboplatin AUC7 in Clinical Stage I Seminomatous Testicular Cancer
Brief Title: Adjuvant Bleomycin, Etoposide and Cisplatin (BEP) Versus Carboplatin in Stage I Seminomatous Testicular Cancer
Acronym: SWENOTECA-ABC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Haukeland University Hospital (Other); University Hospital of North Norway (Other); Sahlgrenska University Hospital (Other); Karolinska Institutet (Other); Oslo University Hospital (Other); Uppsala University Hospital (Other); University Hospital, Linkoeping (Other); Skane University Hospital (Other); Norrlands University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/2012; 2014-004075-23 (EudraCT Number)
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Testicular Neoplasms; Seminoma
Keywords: Chemotherapy, adjuvant; Recurrence; Carboplatin; Bleomycin; Etoposide; Cisplatin
MeSH Terms: conditions — Testicular Neoplasms; Seminoma; Recurrence | interventions — Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bleomycin-Etoposide-Cisplatin (Experimental): One course of adjuvant BEP.
  Interventions: Drug: Bleomycin Etoposide and Cisplatin
- Carboplatin (Active Comparator): One course of adjuvant carboplatin AUC7
  Interventions: Drug: Carboplatin

INTERVENTIONS:
Drug: Bleomycin Etoposide and Cisplatin
  Other Names: BEP
  Arms: Bleomycin-Etoposide-Cisplatin
Drug: Carboplatin
  Other Names: Carboplatin AUC7
  Arms: Carboplatin

SUMMARY:
One course of adjuvant carboplatin AUC7 is considered internationally to be a standard treatment option in clinical stage I seminoma, regardless of risk factors. Treatment is based on a large, randomized phase III study comparing adjuvant carboplatin with adjuvant radiotherapy. This study was done without registering data on possible risk factor for relapse. The relapse rate following carboplatin was in this study estimated to be 5.3 %. Data from a prospective, risk-adapted Spanish study showed that patients without risk factors had a very low risk of relapse, even without adjuvant treatment. This result is also confirmed by a recent analysis of SWENOTECA VII data, showing that this group of patients has a risk of relapse of less than 5 % without adjuvant treatment.

Combined data from SWENOTECA V and VII studies indicate a high risk of relapse in patients with one or two risk factors (tumor 4 cm, stromal invasion of rete testis) treated with one course of adjuvant carboplatin. The relapse rate in this group of patients was 9.4 %, indicating a very modest effect of one course of adjuvant carboplatin. If adjuvant chemotherapy is the preferred treatment strategy, more potent chemotherapy regimens should be explored in this patient group. The results from SWENOTECA III/VI studies with one course of cisplatin-based adjuvant chemotherapy in clinical stage I nonseminoma, show a very low rate of relapse. As seminoma is even more chemosensitive than nonseminoma the relapse rate following one course of adjuvant BEP is expected to be very low, close to 1 %.

The overall aim is to investigate whether one course of adjuvant BEP have a lower relapse rate than one course of adjuvant carboplatin AUC7. In addition, it will be investigated if there is a difference in health related quality of life as well as acute and long-term toxicities from treatment.

DETAILED DESCRIPTION:
Short term overall survival is, regardless of treatment allocation, expected to be very close to 100 %. The primary outcome is relapse rate. The power of the study depends on the number of observed relapses. If the relapse rate in the adjuvant carboplatin group, the reference group, is lower than the anticipated 9 %, we need to include more patients to the study. Based on all previous published material on adjuvant treatment in clinical stage I seminoma it is not possible to precisely estimate the correct relapse rate until the median follow-up is four years. Consequently, we will estimate the relapse rate in the reference group close to the end of accrual. If the estimated relapse rate, and thus the number of relapses, is lower than the anticipated we will increase the sample size to make sure that the study meets the minimum required number of relapses in the reference group. A possible inclusion of more study participants does not compromise the Type I error rate of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of unilateral seminoma testicular cancer, evaluating both size of tumor and invasion of the rete testis
* Clinical stage I
* Tumor size over 4 cm and/or stromal invasion of the rete testis by tumor cells
* Normal value of alpha-fetoprotein (AFP) before orchiectomy. A stable, slightly elevated AFP as a normal value may be permitted.
* Age ≥ 18 years and < 60 years
* Adequate organ function defined as:

Serum aspartate transaminase (ALT) ≤ 1.5 x upper limit of normal (ULN). Total serum bilirubin ≤ 1.5 x ULN Absolute neutrophil count (ANC) ≥ 1.5 x 109/L Platelets ≥ 100 x 109/L Creatinine clearance > 50 ml/min (eGFR) All fertile patients should use safe contraception Written informed consent

Exclusion Criteria:

* Signs of metastatic disease evaluated by CT thorax, abdomen and pelvis. Patients in need of restaging (see SWENOTECA IX) should not be included
* Prior diagnosis of testicular cancer
* Chronic pulmonary disorders giving a high risk of bleomycin induced toxicity (for example chronic obstructive pulmonary disease or lung fibrosis)
* Cancer other than seminoma testicular cancer
* Known hypersensitivity or contraindications for the study drugs
* Serious concomitant systemic disorders (for example active infection, unstable cardiovascular disease) that in the opinion of the investigator would compromise the patient's ability to complete the study or interfere with the evaluation of the efficacy and safety of the study treatment
* Medical, social, psychological conditions that could prevent adequate information and follow-up

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 348 (Estimated)
Dates: Start 2015-04-08 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
Relapse rate | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Olof Ståhl, Md PhD, Principal Investigator — Skane University Hospital; Torgrim Tandstad, MD PhD, Principal Investigator — St. Olavs University Hospital
Locations (2):
- Norway (2):
  - Institutt for kreftforskning og molekylær medisin, St Olavs Hospital, Trondheim
  - St. Olavs University hospital HF, Trondheim